CLINICAL TRIAL: NCT06492057
Title: ElectroMyoStimulation (EMS Body Suit) Protocol to Improve Exercise Outcome in Space Missions (EasyMotion-2)
Brief Title: Electromyostimulation (EMS) of Astronauts in Spaceflight (Easymotion-2)
Acronym: Easymotion-2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: German Sport University, Cologne (Other)
Responsible Party: Principal Investigator, Dieter Blottner, Professor Dr. (PhD), Charite University, Berlin, Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 50WB2329
Record Dates: First submitted 2024-05-23; First posted 2024-07-09 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Muscle Atrophy; Myotonia; Stiffness; Spine; Exercise Overtraining
Keywords: skeletal muscle; passive muscle stiffness; muscle health; electromyostimulation; space flight; countermeasure
MeSH Terms: conditions — Muscular Atrophy; Myotonia; Overtraining Syndrome | interventions — Electromyography; Magnetic Resonance Imaging; Postmortem Imaging

STUDY DESIGN:
Intervention Model Description: In the second phase of their long-duration flight (>130 days or more), each participant wears a personalized Easymotionskin body suit (muscle stimulation suit) controlled by Easymotion App software on crew iPad for only for about 15-20 minutes while performing routine inflight exercise using standard inflight countermeasure devices (treadmill=T2, Cycle Ergometer on ISS, CEVIS; advanced Resistive Exercise Device, ARED) available onboard the ISS. Total EMS exercise time and duration: 12 times EMS plus T2, CEVIS or ARED within 3 weeks on ISS.
Masking Description: Subject A to K
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- EMS (electromyostimulation) participants (Experimental): Healthy Astronauts that perform EMS-assisted inflight exercise onboard the International Space Station
  Interventions: Device: Electromyostimulation (EMS); Device: Myoton; Diagnostic Test: Electromyography (EMG); Diagnostic Test: Magnetic Resonance Imaging (MRI); Diagnostic Test: Dynamometry

INTERVENTIONS:
Device: Electromyostimulation (EMS) — EasymotionSkin body suit for digitally controlled electric impulses via Easymotion-2 software on crew iPad (frequency, impulse rate, duration) are transferred from integrated dry electrodes of the EMS- stimulation suit to activate surface muscle groups of the body (trunk), arms and legs
  Other Names: EMS body muscle stimulation
Device: Myoton — The non-invasive Myoton technology collects data from passive muscle properties (tone and stiffness) obtained from selected anatomical surface muscle groups
  Other Names: passive muscle properties
Diagnostic Test: Electromyography (EMG) — As a standard method, surface EMG collects data from nerve impulse-triggered active muscle contractions, pre/postflight only
  Other Names: surface EMG/nerve impulse rate [amplitude/frequency]
Diagnostic Test: Magnetic Resonance Imaging (MRI) — MRI is a clinically standard (non-radiation) imaging method to study structural changes of the human body (organs, muscle, bones, tendons) at the macroscopic level, pre/postflight only
  Other Names: MRI; Magnetic Resonance Tomography
Diagnostic Test: Dynamometry — Dynamometry is a standard functional and diagnostic method to test muscle strength in sports and rehabilitation. pre/postflight only
  Other Names: muscle functional test

SUMMARY:
This is a prospective spaceflight study involving an investigational non-risk device called the EasyMotionSkin for whole body electric muscle (myo) stimulation (WB-EMS) onboard the International Space Station (ISS).

The purpose of this study is to show:

* optimized exercise outcome with EMS in human spaceflight
* demonstrate efficacy of EMS as alternative inflight exercise protocol
* provide a time-saving and reliable EMS-assisted exercise protocol compliant to astronauts for later use in planetary habitats and future deep space exploration

Eight (n=8) astronauts on long duration missions will take part in this study. This experiment uses the following hardware/software (HW & SW): (A) EasymotionSkin suit (dry electrode muscle stimulation), B) non-invasive hand-held Myoton device (digitized passive muscle stiffness data collection). C) a customized Myoton body template suit (elastic yoga suit with customized anatomical reference labels to aid inflight Myoton data collection on dedicated perforated 2x2 cm small skin fields) at 5 different skin measurement points (MP), neck, back, shoulder, legs.

Before and after flight the following tests will be done once: Myoton data collection, dynamometry strength test, magnetic resonance imaging (MRI) for baseline comparison. Researchers will compare data from a non EMS control group (non EMS Astronauts, retrospective) to see if changes of passive muscle stiffness is seen in EMS Astronauts before, during and after spaceflight

DETAILED DESCRIPTION:
In a previous space analog study (60 days reactive jumps on a sledge during bed rest immobilisation, Cologne, Germany, 2015) on n=24 voluntary participants followed by an experiment on the International Space Station, ISS (MYOTONES 2015-2023) the investigators used non-invasive Myoton technology (Myoton device) to detect digital biomarkers (passive muscle tone and stiffness) on twelve (n=12) study participants together with clinical imaging (MRI), muscle strength tests (dynamometry), and blood samples (biosamples) to study muscle properties and adaptation in microgravity following routine inflight exercise in ISS Astronauts. One of the MYOTONES ISS Astronaut already tested a space-qualified EasymotionSkin suit (Demo-Tech Experiment, German Aerospace Agency, Deutsches Zentrum fuer Luft- und Raumfahrt, DLR, 2022) that was used for about 20 minutes on top of the daily routine exercise protocol in order to optimize inflight training outcome by EMS technology in spaceflight. Preliminary results (n=1) showed feasibility of the novel EMS technology in spaceflight and suggested improved muscle health parameters (increased tone and stiffness) found in some muscle from torso (lower back) and limbs compared to a non-EMS mission crewmember. Easymotion-2 is designed to replicate similar changes in inflight passive muscle parameters (resembling muscle health) in eight (n=8) more ISS Astronauts for robust statistical analyses and interpretation. Pre and postflight baseline data collections with Myoton technology (passive tone [Hz] and stiffness [N/m]) serve as control for comparison. Protocol and recruitment of healthy study participants (male or female Astronauts) is under control by NASA via Informed Consent Briefing standardized procedures.

ELIGIBILITY:
Inclusion Criteria:

Astronauts with active Flight Medical

Exclusion Criteria:

* Heart disease
* Liver disease
* Diabetes
* Thrombosis
* Extreme blood pressure
* Abdominal & inguinal hernias (bulges)
* Strong neurological diseases
* Pregnancy
* Cancer

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Myoton Tone (baseline preflight) | L-105+/-30 days (time window)
  Passive muscle tone [Hz] numerical indices. Abbreviations for Outcome Measures 1-37: Hertz, Hz; Newton/meter, N/m; before launch (preflight), L-; recovery (postflight), R+; inflight days, FD; not earlier than, NET; not later than, NLT; electro-myo-stimulation, EMS; versus/against, vs; surface electromyography, sEMG.
Myoton Tone (recovery postflight) | R+30+/-10 days (time window)
  Passive muscle tone [Hz] numerical indices. Abbreviations for Outcome Measures 1-37: Hertz, Hz; Newton/meter, N/m; before launch (preflight), L-; recovery (postflight), R+; inflight days, FD; not earlier than, NET; not later than, NLT; electromyostimulation, EMS; versus/against, vs; surface electromyography, sEMG.
Myoton Tone (inflight, preEMS-1) | FD20-30 days (time window)
  Passive muscle tone [Hz] numerical indices. Abbreviations: see Outcome1
Myoton Tone (inflight, preEMS-2) | FD60-80 days (time window)
  Passive muscle tone [Hz] numerical indices. Abbreviations: see Outcome1
Myoton Tone (inflight, post EMS-1) | NET R-18 days (time window)
  Passive muscle tone [Hz] numerical indices. Abbreviations: see Outcome1
Myoton Tone (inflight, post EMS-2) | NLT R-12 days (time window)
  Passive muscle tone [Hz] numerical indices. Abbreviations: see Outcome1
Myoton stiffness (baseline, preflight). | L-105+/-30 days (time window)
  Passive muscle stiffness [N/m] numerical indices. Abbreviations: see Outcome 1
Myoton stiffness (recovery, postflight). | R+30+/-10 days (time window)
  Passive muscle stiffness [N/m] numerical indices. Abbreviations: see Outcome 1
Myoton stiffness (inflight, preEMS-1) | FD20-30 days (time window)
  Passive muscle stiffness [N/m] numerical indices. Abbreviations: see Outcome 1
Myoton stiffness (inflight, preEMS-2) | FD60-80 days (time window)
  Passive muscle stiffness [N/m] numerical indices. Abbreviations: see Outcome 1
Myoton stiffness (inflight, postEMS-1) | NET R-18 days (time window)
  Passive muscle stiffness [N/m] numerical indices. Abbreviations: see Outcome 1
Myoton stiffness (inflight, postEMS-2) | NLT R-12 days (time window)
  Passive muscle stiffness [N/m] numerical indices. Abbreviations: see Outcome 1
EMS body stimulation (inflight EMS1) | NET R-60 and NLT R-21 days (time window)
  1st out of a total of 12 (1/12) single EMS-assisted inflight exercise between NET R-60 and NLT R-21 days (time window) with 1-4 days in between "wash-out") at tolerable stimulation merged to nominal daily inflight exercise countermeasure sessions at crew discretion. Applies to Outcome Measures 13-24. Abbreviations: see Outcome 1.
EMS body stimulation (inflight EMS2) | NET R-60 and NLT R-21 days (time window)
  2/12 single EMS-assisted inflight exercise NET R-60 and NLT R-21 days (time window) with 1-4 days in between "wash-out") at tolerable stimulation merged to nominal daily inflight exercise countermeasure sessions at crew discretion. Applies to Outcome Measures 13-24: Abbreviations see Outcome 1.
EMS body stimulation (inflight EMS3) | NET R-60 and NLT R-21 days(time window)
  3/12 single EMS-assisted inflight exercise, NET R-60 and NLT R-21 days (time window) with 1-4 days in between "wash-out")at tolerable stimulation merged to nominal daily inflight exercise countermeasure sessions at crew discretion. Applies to Outcome Measures 13-24: Abbreviations see Outcome 1.
EMS body stimulation (inflight EMS4) | NET R-60 and NLT R-21 days (time window)
  4/12 single EMS-assisted inflight exercise NET R-60 and NLT R-21 days (time window) with 1-4 days in between "wash-out")at tolerable stimulation merged to nominal daily inflight exercise countermeasure sessions at crew discretion. Applies to Outcome Measures 13-24: Abbreviations see Outcome 1.
EMS body stimulation (inflight EMS5) | NET R-60 and NLT R-21 days (time window)
  5/12 single EMS-assisted inflight exercise NET R-60 and NLT R-21 days (time window) with 1-4 days in between "wash-out")at tolerable stimulation merged to nominal daily inflight exercise countermeasure sessions at crew discretion. Applies to Outcome Measures 13-24: Abbreviations see Outcome 1.
EMS body stimulation (inflight EMS6) | NET R-60 and NLT R-21 days (time window)
  6/12 single EMS-assisted inflight exercise NET R-60 and NLT R-21 days (time window) with 1-4 days in between "wash-out")at tolerable stimulation merged to nominal daily inflight exercise countermeasure sessions at crew discretion. Applies to Outcome Measures 13-24: Abbreviations see Outcome 1.
EMS body stimulation (inflight EMS7) | NET R-60 and NLT R-21 days (time window)
  7/12 single EMS-assisted inflight exercise, NET R-60 and NLT R-21 days (time window) with 1-4 days in between "wash-out")at tolerable stimulation merged to nominal daily inflight exercise countermeasure sessions at crew discretion. Applies to Outcome Measures 13-24: Abbreviations see Outcome 1.
EMS body stimulation (inflight EMS8) | NET R-60 and NLT R-21 days (time window)
  8/12 single EMS-assisted inflight exercise NET R-60 and NLT R-21 days (time window) with 1-4 days in between "wash-out") at tolerable stimulation merged to nominal daily inflight exercise countermeasure sessions at crew discretion. Applies to Outcome Measures 13-24: Abbreviations see Outcome 1.
EMS body stimulation (inflight EMS9) | NET R-60 and NLT R-21 days (time window)
  9/12 single EMS-assisted inflight exercise NET R-60 and NLT R-21 days (time window) with 1-4 days in between "wash-out") at tolerable stimulation merged to nominal daily inflight exercise countermeasure sessions at crew discretion. Applies to Outcome Measures 13-24: Abbreviations see Outcome 1.
EMS body stimulation (inflight EMS10) | NET R-60 and NLT R-21 days (time window)
  10/12 single EMS-assisted inflight exercise NET R-60 and NLT R-21 days (time window) with 1-4 days in between "wash-out") at tolerable stimulation merged to nominal daily inflight exercise countermeasure sessions at crew discretion. Applies to Outcome Measures 13-24: Abbreviations see Outcome 1.
EMS body stimulation (inflight EMS11) | NET R-60 and NLT R-21 days (time window)
  11/12 single EMS-assisted inflight exercise NET R-60 and NLT R-21 days (time window) with 1-4 days in between "wash-out") at tolerable stimulation merged to nominal daily inflight exercise countermeasure sessions at crew discretion. Applies to Outcome Measures 13-24: Abbreviations see Outcome 1.
EMS body stimulation (inflight EMS12) | NET R-60 and NLT R-21 days (time window)
  Last out of a total of twelve (12/12) single EMS-assisted inflight exercise NET R-60 and NLT R-21 days (time window) with 1-4 days in between "wash-out") at tolerable stimulation merged to nominal daily inflight exercise countermeasure sessions at crew discretion. Applies to Outcome Measures 13-24: Abbreviations see Outcome 1.
Dynamometry (baseline, preflight/power). | L-105+/-30 days (time window)
  Standard muscle isometric/isokinetic tests (power [Watt] on calf muscle (gastrocnemius) and lower deep back muscle (erector spinae/multifidus). Abbreviations: see Outcome 1
Dynamometry (baseline, preflight/torque). | L-105+/-30 days (time window)
  Standard muscle isometric/isokinetic tests ( torque [Nm]) on calf muscle (gastrocnemius) and lower deep back muscle (erector spinae/multifidus). Abbreviations: see Outcome 1
sEMG (baseline, preflight/amplitude). | L-105+/-30 days (time window)
  Non-invasive sEMG by amplitude on calf muscle (gastrocnemius) and lower deep back muscle (erector spinae/multifidus) as part of dynamometry. Abbreviations: see Outcome 1
sEMG (baseline, preflight/frequency). | L-105+/-30 days (time window)
  Non-invasive sEMG by frequency (Hz) on calf muscle (gastrocnemius) and lower deep back muscle (erector spinae/multifidus) as part of dynamometry. Abbreviations: see Outcome 1
Dynamometry (recovery postflight/power). | R+30+/-10 days (time window)
  Standard muscle isometric/isokinetic tests (power [Watt] on calf muscle (gastrocnemius) and lower deep back muscle (erector spinae/multifidus). Abbreviations: see Outcome 1
Dynamometry (recovery postflight/torque). | R+30+/-10 days (time window)
  Standard muscle isometric/isokinetic tests (torque [Nm] on calf muscle (gastrocnemius) and lower deep back muscle (erector spinae/multifidus). Abbreviations: see Outcome 1
sEMG (recovery postflight/amplitude). | R+30+/-10 days (time window)
  Non-invasive surface EMG (amplitude) on calf muscle (gastrocnemius) and lower deep back muscle (erector spinae/multifidus) as part of dynamometry. Abbreviations: see Outcome 1
sEMG (recovery postflight/frequency). | R+30+/-10 days (time window)
  Non-invasive surface EMG (Hz) on calf muscle (gastrocnemius) and lower deep back muscle (erector spinae/multifidus) as part of dynamometry. Abbreviations: see Outcome 1
Magnetic Resonance Imaging (MRI) (baseline preflight). | L-105+/-30 days (time window)
  Standard clinical structural analysis by optical sections of lower leg and lumbar back muscle profile/volume area (square/3-D, centimeters). Abbreviations: see Outcome 1
Magnetic Resonance Imaging (MRI) (recovery postflight). | R+30+/-10 days (time window)
  Standard clinical structural analysis by optical sections of lower leg and lumbar back muscle profile/volume area (square/3-D, centimeters). Abbreviations: see Outcome 1
EMS protocol report (ms) | NET R-60 and NLT R-21 days (time window)
  Multiple measurements (milliseconds=ms) will be aggregated for each of the 12 single inflight EMS session (see Outcome 13-24) to report on inflight EMS protocol and to collect technical data (of muscle stimulation) for whole body inflight EMS monitoring and assessment. see Outcome1
EMS protocol report (minutes) | NET R-60 and NLT R-21 days (time window)
  Multiple measurements (duration/min.) will be aggregated for each of the 12 single inflight EMS session (see Outcome 13-24) to report on inflight EMS protocol and to collect technical data (of muscle stimulation) for whole body inflight EMS monitoring and assessment. Abbreviations: see Outcome1
EMS protocol report (Hz) | NET R-60 and NLT R-21 days (time window)
  Multiple measurements (frequency/Hz) will be aggregated for each of the 12 single inflight EMS session (see Outcome 13-24) to report on inflight EMS protocol and to collect technical data (of muscle stimulation) for whole body inflight EMS monitoring and assessment. Abbreviations: see Outcome1

CONTACTS AND LOCATIONS:
Overall Officials: Dieter Blottner, PhD, Principal Investigator — Charite-Universitätsmedizin Berlin, Germany
Locations (1):
- Charité - Universitätsmedizin Berlin, Mitte, State of Berlin, Germany

IPD SHARING:
Plan to Share IPD: No
Results will not be shared to other researchers due to privacy reasons of participating Astronauts related to their Space Agencies

REFERENCES:
- [Background] Schoenrock B, Muckelt PE, Hastermann M, Albracht K, MacGregor R, Martin D, Gunga HC, Salanova M, Stokes MJ, Warner MB, Blottner D. Muscle stiffness indicating mission crew health in space. Sci Rep. 2024 Feb 20;14(1):4196. doi: 10.1038/s41598-024-54759-6. PMID 38378866
- [Background] Muckelt PE, Warner MB, Cheliotis-James T, Muckelt R, Hastermann M, Schoenrock B, Martin D, MacGregor R, Blottner D, Stokes M. Protocol and reference values for minimal detectable change of MyotonPRO and ultrasound imaging measurements of muscle and subcutaneous tissue. Sci Rep. 2022 Aug 11;12(1):13654. doi: 10.1038/s41598-022-17507-2. PMID 35953503
- [Background] Schoenrock B, Zander V, Dern S, Limper U, Mulder E, Veraksits A, Viir R, Kramer A, Stokes MJ, Salanova M, Peipsi A, Blottner D. Bed Rest, Exercise Countermeasure and Reconditioning Effects on the Human Resting Muscle Tone System. Front Physiol. 2018 Jul 3;9:810. doi: 10.3389/fphys.2018.00810. eCollection 2018. PMID 30018567

DOCUMENTS (1):
  • Informed Consent Form (2024-01-24): https://cdn.clinicaltrials.gov/large-docs/57/NCT06492057/ICF_000.pdf